CLINICAL TRIAL: NCT04506567
Title: Phase I/II Dose-escalation Study of Fractionated and Multiple Dose 225Ac-J591 for Progressive Metastatic Castration Resistant Prostate Cancer
Brief Title: Fractionated and Multiple Dose 225Ac-J591 for Progressive mCRPC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01021288
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: In schema 1 (dose-fractionated cohort), subject enrollment will be done in a fractionated dose-escalation study design at each dose level with treatment during one cycle to be administered on Day 1 and Day 15.
  In schema 2 (multiple dose cohort), subject enrollment will be done in a dose-escalation single dose study design at each dose level with treatment administered as a single dose per cycle every 6 weeks up to 4 cycles. Additional patients will be enrolled at lower doses previously shown to have efficacy (cohorts -1 and -2). The rationale for enrollment of patients at these lower dosing cohorts is to determine whether a smaller number of cycles at higher radioactivity is superior, inferior, or no different than a larger number of cycles at a lower dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose- Fractionated Cohort (Experimental): Patients will receive a single cycle of 225Ac-J591, administered as a fractionated dose on days 1 and 15. This is a dose-escalation design, with up to 4 dosing cohorts.
  Interventions: Drug: 225Ac-J591; Diagnostic Test: 68Ga-PSMA-HBED-CC injection
- Multiple Dose Cohort (Experimental): Patients will receive 225Ac-J591 every 6 weeks, with up to 4 doses. Some patients will be enrolled in a dose-escalation design, with up to 3 dosing cohorts. Additional patients will be enrolled at 2 lower dosing-cohorts.
  Interventions: Diagnostic Test: 68Ga-PSMA-HBED-CC injection; Drug: 225Ac-J591

INTERVENTIONS:
Drug: 225Ac-J591 — Single cycle of fractionated dose of 225Ac-J591
  Arms: Dose- Fractionated Cohort
Diagnostic Test: 68Ga-PSMA-HBED-CC injection — 68Ga-PSMA-HBED-CC PET/CT before and after treatment
  Other Names: 68Ga-PSMA-11
Drug: 225Ac-J591 — Single dose of 225Ac-J591 every 6 weeks x 4
  Arms: Multiple Dose Cohort

SUMMARY:
The purpose of the initial (phase I) portion of this study is to find a dose level and administration schedule of the study drug, 225Ac-J591, that can be given without severe side effects. The purpose of the second (phase II) portion of the study is to determine the proportion of those with PSMA-positive tumors with >50% PSA decline following 225Ac-J591 treatment in two regimens.

DETAILED DESCRIPTION:
This clinical trial is for men with progressive metastatic castration resistant prostate cancer. The purpose of this study is to find the highest dose level of the study drug, 225Ac-J591, that can be given without severe side effects. The research study is being done because the standard treatments for prostate cancer that has spread beyond the prostate gland are intended to minimize the adverse effects of the disease. These treatments, however, are not curative. Patients who choose to participate in this study will have a screening visit to determine whether or not they are eligible to participate in the study. The treatment phase is comprised of 8 weeks for the fractionated dose cohort (starting from cycle 1, day 1). For the multiple-dose cohort, the dose-limiting toxicity evaluation period is from date of first treatment through treatment on cycle 3, day 1. Following treatment, short-term follow up is planned until radiographic progression, expected to be 6 months.The study medication is called 225Ac-J591, and will be administered as a single fractionated cycle day 1 and day 15 in the fractionated dose regimen and as a single dose per cycle repeated every 6 weeks in the multiple dose regimen. Upon completion of investigational treatment with 225Ac-J591, subjects will undergo 68Ga-PSMA-HBED-CC injection and same day PET/CT at the end of study visit to document treatment response. 68Ga-PSMA-HBED-CC is comprised of gallium-68, which is a positron-emitting radionuclide linked to PSMA-HBED-CC (aka PSMA11), which is a small molecule targeting PSMA. 68Ga-PSMA-HBED-CC will be administered intravenously prior to PET/CT at screening and at follow up imaging x2. Subsequent survival data and additional treatment(s) information will be captured from their routine standard of care (SOC) visits. During the other study visits, participants will undergo routine tests and procedures, such as physical examinations, and blood tests. Some blood tests will be done for research purposes only. After completion of therapy, participants may be contacted on a periodic basis to see how they are doing.

Key eligibility:

* Open to men age 18 and older.
* Diagnosis of progressive metastatic prostate cancer
* Have been previously treated for their disease with particular types of therapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on Prostate Cancer Working

   Group 3 (PCWG3) criteria, which includes at least one of the following criteria:
   * PSA progression
   * Objective radiographic progression in soft tissue
   * New bone lesions
3. Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone orchiectomy
4. Have previously been treated with at least one of the following in any disease state:

   * Androgen receptor signaling inhibitor (such as enzalutamide)
   * CYP 17 inhibitor (such as abiraterone acetate)
5. Have previously received taxane chemotherapy (in any disease state), been determined to be ineligible for taxane chemotherapy by their physician, or refused taxane chemotherapy.
6. Age > 18 years
7. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count >2,000 cells/mm3
   * Hemoglobin ≥9 g/dL
   * Platelet count >150,000 x 109/uL
   * Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault
   * Serum total bilirubin <1.5 x ULN (unless due to Gilbert's Syndrome in which case direct bilirubin must be normal)
   * Serum AST and ALT <3 x ULN in absence of liver metastases; < 5x ULN if due to liver metastases (in both circumstances bilirubin must meet entry criteria)
8. ECOG performance status of 0-2
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

1. Implantation of investigational medical device ≤4 weeks of Treatment Visit 1 (Day 1) or current enrollment in oncologic investigational drug or device study
2. Use of investigational drugs ≤4 weeks or <5 half-lives of Cycle 1, Day 1 or current enrollment in investigational oncology drug or device study
3. Prior systemic beta-emitting bone-seeking radioisotopes
4. Known active brain metastases or leptomeningeal disease
5. History of deep vein thrombosis and/or pulmonary embolus within 1 month of C1D1
6. Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
7. Radiation therapy for treatment of PC ≤4 weeks of Day 1 Cycle 1
8. Patients on stable dose of bisphosphonates or denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the DLT-assessment period of the study
9. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 month after last study drug administration
10. Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse
11. Known history of myelodysplastic syndrome

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male patients of >18 years age with documented progressive metastatic CRPC
Enrollment: 60 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicity (DLT) | Will be collected from Day 1 through 6 months
  DLTs will be measured by utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Cumulative maximum tolerated dose (MTD) | Will be collected from Day 1 through 6 months
  The dose that produces an "acceptable" level of toxicity or that, if exceeded, would put subjects at "unacceptable" risk for toxicity. MTD is defined as the dose level at which no more than two patients out of six experienced dose-limiting toxicity (DLT).
Assess the recommended phase II dose (RP2D) of 225Ac-J591 in fractionated dose and multiple dose regimens (phase I) | Will be collected from Day 1 through 6 months
Assess the proportion of those with PSMA+ tumors with >50% PSA decline following 225Ac-J591 in two regimens (phase II) | Will be collected from Day 1 through 6 months
  Proportion of patients achieving 50% or greater PSA decline (relative to baseline/pre-treatment PSA). Response may occur at any time following treatment initiation and prior to going off study or initiation of new therapy.

SECONDARY OUTCOMES:
Number of subjects with radiographic response | Imaging performed at timepoints from Day 1 through study completion up to 3 years
  Response evaluation criteria in solid tumors RECIST (Version 1.1) criteria with prostate cancer working group 3 (PCWG3) modifications will be used
Overall survival following fractionated dose and multiple doses of 225Ac-J591 | Survival will be collected from Day 1 through study completion up to 3 years
  Overall survival will be captured through in-clinic or telephone contact with subjects
Change in disease assessment with 68Ga-PSMA-11 PET/CT prior to and following investigational treatment | Scans will be performed at screening, day 85 and day 168
  68Ga-PSMA-11 PET/CT will be utilized as part of the radiographic assessment.
Change in circulating tumor cells (CTC) and the rate of favorable and undetectable CTC count at 12 weeks following 225Ac-J591 | Samples will be collected at screening, day 1, day 85 and at disease progression
  CTCs will be analyzed through blood specimen collection via CellSearch methodology lab testing
Safety of treatment and adverse event rate | Will be collected from Day 1 through study completion up to 3 years
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 is used to grade all adverse events
Assess biochemical progression-free survival | Will be collected from Day 1 through study completion up to 3 years
  PSA progression will be defined as a rise of > 25% above either the pretreatment level or the nadir PSA level (whichever is lowest). PSA must increase by > 2 ng/ml to be considered progression
Assess the proportion with different levels of PSA decline following 225Ac-J591 | Will be collected from Day 1 through study completion up to 3 years
  PSA will be monitored through serial blood draws. Response may occur at any time following treatment initiation and prior to going off study or initiation of new therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Osborne, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Brooklyn Methodist Hospital - New York Presbyterian, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No